CLINICAL TRIAL: NCT04260984
Title: Effect of Ultrasound-guided Corticosteroid Injection Versus Palpation-guided Injection for de Quervain's Disease: a Randomized Control Trial
Brief Title: Effect of Ultrasound-guided Corticosteroid Injection Versus Palpation-guided Injection for de Quervain's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lin-Fen Hsieh, Principal Investigator, Shin Kong Wu Ho-Su Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190705R; 2020SKHADR036 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2020-01-20; First posted 2020-02-07 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: De Quervain Disease
Keywords: De Quervain Disease; ultrasound-guided injection; intra-articular injection
MeSH Terms: conditions — De Quervain Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palpation-guided injection (Active Comparator): Injectate: a mixture of 10mg triamcinolone acetonide (10mg/1ml) and 0.3ml 1% lidocaine. For palpation-guided injection, a 2.5cm 25-gauge needle will be inserted almost horizontally between APL and EPB tendons, just distal to the radial styloid, at the site of maximum tenderness. Then the mixture of triamcinolone and lidocaine will be pushed into the common tendon sheath.
  Interventions: Procedure: palpation-guided injection
- US-guided injection (Active Comparator): For US-guided injection, a 22 MHZ linear array probe (Esaote MyLab™ClassC, Italy) will be used for guidance of injection via a transverse scan, in-plane approach. After sterilization, the probe will be placed at the radial styloid with maximal swelling or tenderness. Then a 2.5 cm 25-gauge needle will be placed into the tendon sheath via transverse scan, in-the-plane approach, and the injectate will be pushed into the tendon sheath. Care will be taken avoiding injury of vessels and the superficial branch of radial nerve during the injection.
  Interventions: Procedure: US-guided injection

INTERVENTIONS:
Procedure: US-guided injection — For US-guided injection, a 22 MHZ linear array probe (Esaote MyLab™ClassC, Italy) will be used for guidance of injection via a transverse scan, in-plane approach. After sterilization, the probe will be placed at the radial styloid with maximal swelling or tenderness. Then a 2.5 cm 25-gauge needle will be placed into the tendon sheath via transverse scan, in-the-plane approach, and the injectate will be pushed into the tendon sheath. Care will be taken avoiding injury of vessels and the superficial branch of radial nerve during the injection.
  Arms: US-guided injection
Procedure: palpation-guided injection — Injectate: a mixture of 10mg triamcinolone acetonide (10mg/1ml) and 0.3ml 1% lidocaine. For palpation-guided injection, a 2.5cm 25-gauge needle will be inserted almost horizontally between APL and EPB tendons, just distal to the radial styloid, at the site of maximum tenderness. Then the mixture of triamcinolone and lidocaine will be pushed into the common tendon sheath.
  Arms: palpation-guided injection

SUMMARY:
The purposes of this study are to compare the effectiveness and side effects of US-guided and palpation-guided corticosteroid injections for de Quervain's disease.

DETAILED DESCRIPTION:
De Quervain's disease is a common clinical disorder, characterized by pain at radial side of the wrist. It often interferes wrist and thumb movement, and may affect activity of daily life. It is caused by overuse and impaired gliding of the abductor pollicis longus (APL) and extensor policis brevis (EPB) tendons at the styloid process of the radius. It is associated with postpartum baby care, or jobs or hobbies that involve repetitive hand and wrist motions. The most effective treatment is corticosteroid injection into the tendon sheath of the conjoined tendons of APL and EPB. Over the past few years because of advancement of sonography in the musculoskeletal system, ultrasound (US)-guided intra-sheath injection has become popular, and it has been proved to improve the accuracy of placement of needle tip in the tendon sheath, however, studies comparing the effect and side effects of US-guided corticosteroid injection with palpation-guided injection for de Quervain's disease have never been reported before. The purposes of this study are to compare the effectiveness and side effects of US-guided and palpation-guided corticosteroid injections for de Quervain's disease.

The investigators plan to recruit 70 patients with de Quervain's disease, half of them will be randomly assigned into US-guided injection group, and the other half into the palpation-guided injection group. Each subject will receive one shot of injection and each subject will expect to fill in the evaluation form at baseline, and at 1 week, 3 months, and 6 months after the injection. Statistics will be performed after completing the patients' treatment and evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Pain and tenderness at the radial side of the wrist.
2. Positive Finkelstein sign, or pain on resistive maximal isometric contraction of extension and/or abduction of the affected thumb.
3. pain intensity on a 10-point visual analog scale (VAS) for pain to ≧ 3 on active thumb abduction or extension.
4. Patient agrees to receive either palpation-guided or US-guided local corticosteroid injection.
5. Age ≧ 20 years old.

Exclusion Criteria:

1. Presence of an absolute contraindication for corticosteroids or local anesthetics injection.
2. During pregnancy.
3. Severe systemic diseases with poor control.
4. Prior treatment with corticosteroid injection and/or surgery at the same anatomical location in the last 6 months.
5. Being unable to fill-in the follow-up forms.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
QuickDASH | 1 week after injection
  QuickDASH is a self-report questionnaire comprising 11 items that focuses on symptoms and the ability to perform certain upper extremity activities on a five-point Likert-type scale. The scores range from 0 (the best) to 100 (the worst). The reliability of QuickDASH was 0.93, and the validity based on response of full-length DASH was 0.96.18

SECONDARY OUTCOMES:
VAS pain | beginning of the treatment and at 1 week ,3 months and 6 months after the beginning of the treatment.
  The patient or the assessor recorded the level of perceived pain by making a vertical mark between the 2 ends of a 10-cm horizontal line. The 0-cm point would represent no pain, while the 10-cm end represents the most extreme pain imaginable. The distance from 0cm to the mark was measured. The reliability of VAS for pain is .94.19
Direct treatment response | beginning of the treatment and at 1 week ,3 months and 6 months after the beginning of the treatment.
  Direct treatment response includes 4 grades: grade 1 is no response, very unsatisfactory; grade 2, partial response, not satisfactory, need further therapy; grade 3, partial response, satisfactory, not warranting further therapy; grade 4, complete symptom relief, very satisfactory.20 Improvement as perceived by patients using a 5-point Likert scale: 1, much worse; 2, worse; 3, same; 4, better; 5, much better.

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No